CLINICAL TRIAL: NCT03715205
Title: A Prospective, Open-label, Phase 4 Study to Evaluate the Safety of Pembrolizumab (KEYTRUDA®) in Subjects With Unresectable or Metastatic Melanoma or PD-L1 Positive Non-small Cell Lung Cancer (NSCLC) in India (Keynote-593)
Brief Title: Study to Evaluate the Safety of Pembrolizumab in Participants With Unresectable or Metastatic Melanoma or Non-small Cell Lung Cancer in India (MK-3475-593/KEYNOTE-593)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-593; MK-3475-593 (Other: MSD); KEYNOTE 593 (Other: MSD)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 200 mg IV Q3W (Experimental): Participants with melanoma or NSCLC receive 200 mg of pembrolizumab as an intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 cycles.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
This study has been designed to evaluate the safety of pembrolizumab in participants in India with unresectable or metastatic melanoma and participants with non-small cell lung cancer (NSCLC) who are either untreated (programmed cell death ligand 1 [PD-L1] ≥50%) or have experienced disease progression after a platinum-containing systemic therapy (PD-L1 ≥1%).

ELIGIBILITY:
Inclusion Criteria:

Melanoma Participant:

* Has a histologically confirmed diagnosis of unresectable Stage III or metastatic melanoma (Stage IV) not amenable to local therapy
* Has received no more than 1 line of prior systemic therapy for unresectable Stage III or Stage IV melanoma including mitogen activated protein kinase inhibitors
* Has a Lactate Dehydrogenase (LDH) ≤1.5 times ULN

NSCLC Participant-First Line Treatment:

* Has a histologically or cytologically confirmed diagnosis of Stage IV NSCLC
* Has a tumor that demonstrate PD-L1 strong expression (PD-L1 ≥50%)
* Do not have an EGFR sensitizing mutation AND are anaplastic lymphoma kinase (ALK) translocation negative
* Has received no systemic anti-cancer therapy for their metastatic NSCLC

NSCLC Participant-Second Line Treatment and Beyond:

* Has a histologically or cytologically confirmed diagnosis of stage IIIB//IIIC/IV (including any future updates to the American Joint Committee on Cancer [AJCC] guideline) or recurrent NSCLC
* Has a tumor that expresses programmed cell death ligand 1 (PD-L1) ≥1%
* Has received prior treatment with at least two cycles of a platinum-containing doublet for Stage IIIB/IV or recurrent disease
* Has received an epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (either erlotinib, gefitinib, or afatinib) if they have an EGFR sensitizing mutation
* Has received crizotinib if they have an ALK translocation

NSCLC participants must also meet the following requirements:

* Have a life expectancy of at ≥3 months
* Provide a formalin fixed tumor tissue sample for PD-L1 biomarker analysis from a recent biopsy of a tumor lesion not previously irradiated; For first line, biopsies obtained PRIOR to the administration of any systemic therapy administered for the treatment of a tumor (such as neoadjuvant/adjuvant/definitive therapy) will not be permitted for analysis. For second line treatment and beyond, no systemic antineoplastic therapy may be administered between the PD-L1 biopsy and initiating study medication
* Have documented evidence of the EGFR mutation status or ALK translocation status. If unable to provide documentation of these molecular changes, formalin-fixed paraffin-embedded tumor tissue of any age should be submitted for testing
* Have measurable disease per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the local site investigator/radiologist
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Women of childbearing potential (WOCP) must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* WOCP must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of trial treatment
* Men of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* For NSCLC Participant only: Has a tumor specimen that is not evaluable for PD-L1 expression by the laboratory
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment
* Has received prior therapy with an anti- programmed cell death 1 (PD-1), anti-PD-L1, or anti- programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another T-cell receptor (i.e., cytotoxic T-lymphocyte antigen-4 [CTLA-4], OX-40, CD137) or has previously participated in a clinical trial for pembrolizumab (MK-3475)
* Has received prior anti-cancer therapy including investigational agent or device within 4 weeks, or completed palliative radiotherapy within 7 days, prior to enrollment
* Has recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline
* Has recovered adequately from the toxicity and/or complications from major surgery prior to starting trial treatment
* Is expected to require any other form of antineoplastic therapy while participating in the trial
* Is on systemic corticosteroid therapy within 7 days before the planned date for first dose of treatment or any other form of immunosuppressive medication
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (exceeding 10 mg daily dose of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a known additional malignancy that is progressing or requires active treatment with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical cancer in situ, breast carcinoma) that have undergone potentially curative therapy
* Has had an allogeneic tissue/solid organ transplant
* Has a history of or current radiographically detectable central nervous system metastases and/or carcinomatous meningitis
* Has a severe hypersensitivity (≥ Grade 3) to any excipients in pembrolizumab
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy including known history of active tuberculosis (Bacillus tuberculosis)
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HbsAg] reactive) or hepatitis C (HCV) ribonucleic acid (RNA) [qualitative] is detected
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
* If participant received prior radiation therapy to a symptomatic metastatic lesion, has recovered to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Grade 1 or Grade 0 AEs due to radiation therapy
* Is a regular user of any illicit drug or has a recent history (within the last 3 months) of substance abuse including alcohol
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received a live vaccine within 30 days before the first dose of trial treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- India (8):
  - Nizam's Institute of Medical Sciences ( Site 0011), Hyderabad, Andhra Pradesh
  - Artemis Health Institute ( Site 0007), Gurgaon, Haryana
  - Tata Memorial Hospital [M] ( Site 0005), Mumbai, Maharashtra
  - Kokilaben Ben Dhirubhai Ambani Hosp & Med Res Inst. ( Site 0001), Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Center ( Site 0009), Pune, Maharashtra
  - All India Institute of Medical Sciences ( Site 0012), New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals ( Site 0008), New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute and Research Centre ( Site 0003), Delhi

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with unresectable or metastatic melanoma, or Non-small Cell Lung Cancer (NSCLC) who were either treatment naïve or had disease progression after prior treatment, were recruited to the study.
Pre-assignment Details: Of 284 participants screened, 150 were allocated to receive pembrolizumab.
Groups:
- Pembrolizumab 200 mg IV Q3W: Participants with melanoma or NSCLC received 200 mg of pembrolizumab as an IV infusion Q3W for up to 35 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg IV Q3W
Started | 150
Completed | 16
Not Completed | 134
Not completed — Death | 13
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 93
Not completed — Withdrawal by Subject | 26

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 150
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 150
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. The number of participants with an AE was reported.
Time Frame: Up to approximately 66.5 months
Population: All participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 131

2. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. An SAE was any adverse event occurring at any dose or during any use of Sponsor's product that resulted in death; was life threatening; resulted in persistent or significant disability/incapacity; resulted in or prolonged an existing inpatient hospitalization; was a congenital anomaly/birth defect; was another important medical event. The number of participants with an SAE was reported.
Time Frame: Up to approximately 66.5 months
Population: All participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 31

3. Primary Outcome: Number of Participants With a Drug-Related AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. A drug-related AE was defined as an AE that was determined by the investigator to be possibly, probably, or definitely related to drug. The number of participants with a drug-related AE was reported.
Time Frame: Up to approximately 66.5 months
Population: All participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 61

4. Primary Outcome: Number of Participants With a Drug-Related SAE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An SAE was any AE occurring at any dose or during any use of Sponsor's product that resulted in death; was life threatening; resulted in persistent or significant disability/incapacity; resulted in or prolonged an existing inpatient hospitalization; was a congenital anomaly/birth defect; was another important medical event. A drug-related SAE was defined as an SAE that was determined by the investigator to be possibly, probably, or definitely related to drug. The number of participants with a drug-related SAE was reported.
Time Frame: Up to approximately 66.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 10

5. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. The number of participants who discontinued study drug due to an AE was reported
Time Frame: Up to approximately 26 months
Population: All participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 11

6. Other Pre Specified Outcome: Number of Participants With an Adverse Event of Special Interest (AEOSI)
Description: An AEOSI was defined as an AE (serious or non-serious) of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor was appropriate. Pembrolizumab AEOSIs included immune-mediated events (pneumonitis, colitis, hepatitis, nephritis, adrenal insufficiency, hypophysitis, hyperthyroidism, hypothyroidism, thyroiditis, type 1 diabetes mellitus, severe skin reactions including Stevens-Johnson Syndrome [SJS] and Toxic Epidermal Necrolysis [TEN], uveitis, pancreatitis, myositis, Guillain-Barre Syndrome, myocarditis, encephalitis, sarcoidosis, myasthenic syndrome, myelitis, vasculitis, cholangitis sclerosing, hypoparathyroidism, arthritis, haemophagocytic lymphohistiocytosis, optic neuritis, gastritis, haemolytic anaemia, exocrine pancreatic insufficiency, pericarditis) and infusion reactions. The number of participants with an AEOSI was reported.
Time Frame: Up to approximately 66.5 months
Population: All participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg IV Q3W
Number analyzed (Participants) | 150
Participants | 33

ADVERSE EVENTS:
Time Frame: Up to approximately 66.5 months
Description: All-Cause Mortality reported for all randomized participants.
  Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab 200 mg IV Q3W
All-Cause Mortality (participants affected / at risk) | 13/150
Serious Adverse Events (participants affected / at risk) | 31/150
Other Adverse Events (participants affected / at risk) | 105/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg IV Q3W (N=150)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg IV Q3W (N=150)
Anaemia (Blood and lymphatic system disorders) | 19 (21)
Hypothyroidism (Endocrine disorders) | 26 (27)
Abdominal pain (Gastrointestinal disorders) | 10 (11)
Constipation (Gastrointestinal disorders) | 17 (18)
Vomiting (Gastrointestinal disorders) | 11 (11)
Asthenia (General disorders) | 8 (8)
Fatigue (General disorders) | 17 (18)
Pyrexia (General disorders) | 15 (26)
Urinary tract infection (Infections and infestations) | 15 (17)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15)
Rash (Skin and subcutaneous tissue disorders) | 9 (10)
Vitiligo (Skin and subcutaneous tissue disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03715205/Prot_SAP_000.pdf